CLINICAL TRIAL: NCT02660840
Title: Interventional, Open-label, Randomised, Crossover, Comparative Study of the Pharmacokinetics and Bioequivalence of Two Flupentixol Formulations - Film Coated Tablet (Test Treatment) - 0.5 mg, 1 mg and 5 mg (H. Lundbeck A/S, Denmark) and Coated Tablet (Fluanxol®) - 0.5 mg, 1 mg and 5 mg (H. Lundbeck A/S, Denmark) in Healthy Volunteers
Brief Title: Comparative Study of the Pharmacokinetics and Bioequivalence of Two Flupentixol Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15969A
Record Dates: First submitted 2016-01-19; First posted 2016-01-21 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Bioequivalence Study in Healthy Subjects
MeSH Terms: interventions — Flupenthixol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 0.5 mg Test, then 0.5 mg reference (Experimental): 14 Subjects will receive a 0.5 mg single dose of two different pharmaceutical formulations (first test, then reference)
  Interventions: Drug: 0.5 mg Flupentixol film-coated tablet (test treatment); Drug: 0.5 mg Flupentixol coated tablet (reference treatment)
- 0.5 mg reference, then 0.5 mg Test (Experimental): 14 Subjects will receive a 0.5 mg single dose of two different pharmaceutical formulations (first reference, then test)
  Interventions: Drug: 0.5 mg Flupentixol film-coated tablet (test treatment); Drug: 0.5 mg Flupentixol coated tablet (reference treatment)
- 1 mg Test, then 1 mg reference (Experimental): 14 Subjects will receive a 1 mg single dose of two different pharmaceutical formulations (first test, then reference)
  Interventions: Drug: 1 mg Flupentixol film-coated tablet (test treatment); Drug: 1 mg Flupentixol coated tablet (reference treatment)
- 1 mg reference, then 1 mg Test (Experimental): 14 Subjects will receive a 1 mg single dose of two different pharmaceutical formulations (first reference, then test)
  Interventions: Drug: 1 mg Flupentixol film-coated tablet (test treatment); Drug: 1 mg Flupentixol coated tablet (reference treatment)
- 5 mg Test, then 5 mg reference (Experimental): 14 Subjects will receive a 5 mg single dose of two different pharmaceutical formulations (first test, then reference)
  Interventions: Drug: 5 mg Flupentixol film-coated tablet (test treatment); Drug: 5 mg Flupentixol coated tablet (reference treatment)
- 5 mg reference, then 5 mg Test (Experimental): 14 Subjects will receive a 5 mg single dose of two different pharmaceutical formulations (first reference, then test)
  Interventions: Drug: 5 mg Flupentixol film-coated tablet (test treatment); Drug: 5 mg Flupentixol coated tablet (reference treatment)

INTERVENTIONS:
Drug: 0.5 mg Flupentixol film-coated tablet (test treatment) — single oral dose, fasted state, day 1 in period 1 or 2
  Arms: 0.5 mg Test, then 0.5 mg reference; 0.5 mg reference, then 0.5 mg Test
Drug: 1 mg Flupentixol film-coated tablet (test treatment) — single oral dose, fasted state, day 1 in period 1 or 2
  Arms: 1 mg Test, then 1 mg reference; 1 mg reference, then 1 mg Test
Drug: 5 mg Flupentixol film-coated tablet (test treatment) — single oral dose, fasted state, day 1 in period 1 or 2
  Arms: 5 mg Test, then 5 mg reference; 5 mg reference, then 5 mg Test
Drug: 0.5 mg Flupentixol coated tablet (reference treatment) — single oral dose, fasted state, day 1 in period 1 or 2
  Other Names: Fluanxol®
  Arms: 0.5 mg Test, then 0.5 mg reference; 0.5 mg reference, then 0.5 mg Test
Drug: 1 mg Flupentixol coated tablet (reference treatment) — single oral dose, fasted state, day 1 in period 1 or 2
  Other Names: Fluanxol®
  Arms: 1 mg Test, then 1 mg reference; 1 mg reference, then 1 mg Test
Drug: 5 mg Flupentixol coated tablet (reference treatment) — single oral dose, fasted state, day 1 in period 1 or 2
  Other Names: Fluanxol®
  Arms: 5 mg Test, then 5 mg reference; 5 mg reference, then 5 mg Test

SUMMARY:
To establish bioequivalence between new film-coated tablet formulations of 0.5 mg, 1 mg and 5 mg flupentixol and the marketed coated tablet formulations of 0.5 mg, 1 mg, and 5 mg flupentixol, administered as single doses

DETAILED DESCRIPTION:
All subjects will be confined to the clinic from Day -1 (Baseline) until Day 6 (120 hours post-dose) for each dosing period. First and second dosing will be separated by a washout period of at least 21 days

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of ≥18.5 and ≤30 kg/m2
* The subject is, in the opinion of the investigator, generally healthy based on medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The subject is pregnant or breastfeeding.
* The subject has taken any investigational medicinal products 3 months prior to the first dose
* The subject has tested positive at the Screening Visit or at the Baseline Visit for drugs of abuse (opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates, benzodiazepines, and cannabinoids).

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve | from 0 to 72 hours post-dose
The maximum observed concentration (Cmax) | from 0 to 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- RU801, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided